CLINICAL TRIAL: NCT02764606
Title: CANPOS: Predictive Biomarkers of Tumor Progression in Non-small Cell Lung Cancer
Acronym: CANPOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50832
Record Dates: First submitted 2016-04-28; First posted 2016-05-06 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer; Biomarkers; Bone; Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a non-small cell lung cancer: Serum and plasma samples (at time of diagnosis, after surgery, and at time of progression to evaluate the value of new serum markers to predict the occurrence of metastases).
  Interventions: Biological: Serum and plasma samples

INTERVENTIONS:
Biological: Serum and plasma samples — Serum and plasma are collected at time of diagnosis, after surgery, and at time of progression to evaluate the value of new serum markers to predict the occurrence of metastases.

SUMMARY:
CANPOS is a non-interventional study aiming at evaluate at the time of initial surgery the value of new serum markers to predict the occurrence of metastases in patients with early-stage non-small cell lung cancer. This would represent a rational to develop personalized follow-up and prevention strategies

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis or suspected for a diagnosis of lung cancer, non-small cell lung cancer
* age over 18 years
* patient naïve of any oncology treatment (excluding surgery alone) within the past 5 years
* patient who signed the informed consent by the study protocol

Exclusion criteria were:

* any ongoing treatment for cancer
* any history of cancer within 5 years before the diagnosis of lung cancer
* any psychological, sociological or geographical conditions that would not allow the study follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early-stage non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Serum levels of osteoprotegerin | At the time of initial surgery
  The serum levels of osteoprotegerin, as assessed by standard ELISA methods, will be measured to to evaluate at the time of initial surgery, the value of new serum markers to predict the occurrence of metastases in patients with early-stage non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon / Hôpital Neurologique Pierre Wertheimer, Bron, France